CLINICAL TRIAL: NCT00185952
Title: Nifedipine for the Maintenance Tocolysis of Preterm Labor: Comparison to Placebo in a Prospective, Randomized Double Blind Trial
Brief Title: Nifedipine vs Placebo for Maintenance Tocolysis of Preterm Labor.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Santa Clara Valley Health & Hospital System (Other)
Responsible Party: Yasser Yehia El-Sayed, Stanford University School of Medicine
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 76251
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2011-06-13 (Estimated); Status verified 2011-06

CONDITIONS: Obstetric Labor, Premature; Venous Thrombosis
MeSH Terms: conditions — Obstetric Labor, Premature; Venous Thrombosis | interventions — Nifedipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nifedipine (Active Comparator): Maintenance tocolysis with nifedipine.
  Interventions: Drug: Nifedipine
- Placebo (Placebo Comparator): Maintenance tocolysis with placebo tablets.
  Interventions: Drug: Nifedipine

INTERVENTIONS:
Drug: Nifedipine — Nifedipine 10 mg tablets, two tablets orally every 6 hours. Placebo tablets, two tablets orally every 6 hours.

SUMMARY:
Comparing nifedipine to placebo for the maintenance tocolysis of preterm labor

DETAILED DESCRIPTION:
To estimate whether maintenance nifedipine tocolysis after arrested preterm labor prolongs pregnancy and improves neonatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

- arrested preterm labor

Exclusion Criteria:

- ruptured membranes, fetal distress, placenta previa, placental abruption, maternal medical contraindication to tocolysis

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2001-11; Primary Completion 2007-01 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Achieving 37 weeks gestation | delivery

SECONDARY OUTCOMES:
Incidence of recurrent preterm labor | Delivery
Neonatal outcomes | Discharge of neonate

CONTACTS AND LOCATIONS:
Overall Officials: Yasser Yehia El-Sayed, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Result] Lyell DJ, Pullen KM, Mannan J, Chitkara U, Druzin ML, Caughey AB, El-Sayed YY. Maintenance nifedipine tocolysis compared with placebo: a randomized controlled trial. Obstet Gynecol. 2008 Dec;112(6):1221-1226. doi: 10.1097/AOG.0b013e31818d8386. PMID 19037029
- [Derived] Wilson A, Hodgetts-Morton VA, Marson EJ, Markland AD, Larkai E, Papadopoulou A, Coomarasamy A, Tobias A, Chou D, Oladapo OT, Price MJ, Morris K, Gallos ID. Tocolytics for delaying preterm birth: a network meta-analysis (0924). Cochrane Database Syst Rev. 2022 Aug 10;8(8):CD014978. doi: 10.1002/14651858.CD014978.pub2. PMID 35947046